CLINICAL TRIAL: NCT03663686
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose, Single-center Study to Assess the Safety, Tolerability and Pharmacokinetic of Litapiprant Tablets in Healthy Subjects
Brief Title: The Safety, Tolerability and Pharmacokinetic Study of Litapiprant Tablets in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC46877-P-01
Record Dates: First submitted 2018-09-02; First posted 2018-09-10 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2018-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 25mg single doses (Placebo Comparator): Intervention Drug: 25mg Litapiprant Tablet administered orally once daily Intervention Drug: Matching Placebo Tablet administered orally once daily
  Interventions: Drug: Litapiprant Tablet
- 50mg single doses (Placebo Comparator): Intervention Drug: 50mg Litapiprant Tablet administered orally once daily Intervention Drug: Matching Placebo Tablet administered orally once daily
  Interventions: Drug: Litapiprant Tablet
- 100mg single doses (Placebo Comparator): Intervention Drug: 100mg Litapiprant Tablet administered orally once daily Intervention Drug: Matching Placebo Tablet administered orally once daily
  Interventions: Drug: Litapiprant Tablet
- 200mg single doses (Placebo Comparator): Intervention Drug: 200mg Litapiprant Tablet administered orally once daily Intervention Drug: Matching Placebo Tablet administered orally once daily
  Interventions: Drug: Litapiprant Tablet
- 400mg single doses (Placebo Comparator): Intervention Drug: 400mg Litapiprant Tablet administered orally once daily Intervention Drug: Matching Placebo Tablet administered orally once daily
  Interventions: Drug: Litapiprant Tablet
- 600mg single doses (Placebo Comparator): Intervention Drug: 600mg Litapiprant Tablet administered orally once daily Intervention Drug: Matching Placebo Tablet administered orally once daily
  Interventions: Drug: Litapiprant Tablet
- 800mg single doses (Placebo Comparator): Intervention Drug: 800mg Litapiprant Tablet administered orally once daily Intervention Drug: Matching Placebo Tablet administered orally once daily
  Interventions: Drug: Litapiprant Tablet

INTERVENTIONS:
Drug: Litapiprant Tablet — Small molecules inhibitors of the chemoattractant receptor homologous molecule expressed on Th2 cells

SUMMARY:
The Safety, Tolerability and Pharmacokinetic Study of Asthma Treatment Drug Litapiprant Tablets in Healthy Male and Female subjects.

DETAILED DESCRIPTION:
This was a Randomized，Double-blind, Placebo-controlled, Single Ascending Dose, Single-center Study to Assess the Safety, Tolerability and Pharmacokinetic of Litapiprant Tablets in Healthy Male and Female subjects. A total of 60 healthy subjects were divided into 7 groups. Group 1 consist of 4 subjects, 3 subjects will receive Litapiprant Tablets and 1 subject will receive placebo.Group 2,3,5,6 consist of 8 subjects respectively, in each group, 6 subjects will receive Litapiprant Tablets and 2 subjects will receive placebo.Group 4,7 consist of 12 subjects respectively, in each group, 10 subjects will receive Litapiprant Tablets and 2 subjects will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, overall healthy subjects，female VS male 1:1 ratio;
* Between 18 and 45 years of age, inclusive, similar ages;
* Body weight should be≥50 kg; Body Mass Index (BMI) is between 19.0 and 28.0 kg/m2, inclusive;
* Able to comprehend and sign the ICF voluntarily prior to initiate the study;
* Able to communicate well with the investigator and complete the study according to the protocol.

Exclusion Criteria:

* Pregnant or nursing female, or plan for pregnancy within 6 months;
* A clinically significant abnormal finding on the physical exam, medical history, electrocardiogram (ECG), or clinical laboratory results at screening;
* Has a positive test for hepatitis B surface antigen, hepatitis C antibody, syphilis antibody， or HIV antibody . A clinically significant abnormal finding on HBV-DNA test ;
* Sitting systolic blood pressure (SBP) <90mmHg or >140mmHg, and/or sitting diastolic blood pressure (DBP) <60mmHg or >90mmHg at screening;
* With the history of using any drug which will inhibit or induce liver metabolize drug and/or will infect gastric acid within 1 month before randomization;
* Receipt of any medication including over the counter preparations and vitamins within 14 days of the first study day;
* History of cardiovascular, immune system, Severe digestive system, Circulatory system, respiratory system, urinary system , nervous system,tumor diseases;
* Suffering from blood diseases such as coagulopathy;
* Patients with a history of mental illness or active mental illness;
* Have undergone major surgery within 6 months before enrollment;
* A history of gastrointestinal, liver ,kidney diseases likely to influence drug absorption within 6 months before enrollment;
* Drug or alcohol abuse;
* History of drug abuse and drug use within 1 year prior to the study;
* Habitual consumption of grapefruit juice, tea, coffee and/or caffeinated beverages, which cannot be withdrawn during the trial;
* The average daily smoking volume is >5 within 3 months prior to the study;
* A history of hypersensitivity and/or idiosyncrasy to any of the test compounds or related drugs or excipients employed in this study;
* Participation in a clinical study within 3 months of the first dose of study drug;
* Donation of blood within 3 months of the first dose of study drug or have a plan to donate blood;
* Cannot be tolerant to oral drugs;
* Poor peripheral venous access conditions;
* The investigator believes that it should not be included;
* Additional exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Adverse events | Baseline to day 8~10
  To assess the safety and tolerability after a single dose of Litapiprant Tablets

SECONDARY OUTCOMES:
AUC0-∞ | Prior to dosing（0 hour）and 0.25 hour、0.5 hour、1 hour、1.5 hours、2 hours、3 hours、4 hours、6 hours、8 hours、10 hours、12 hours、24 hours、36 hours、48 hours、72 hours、96 hours after dosing
  area under the concentration versus time curve (AUC) from time zero to infinity
AUC0-t | Prior to dosing（0 hour）and 0.25 hour、0.5 hour、1 hour、1.5 hours、2 hours、3 hours、4 hours、6 hours、8 hours、10 hours、12 hours、24 hours、36 hours、48 hours、72 hours、96 hours after dosing
  AUC from time zero to the time of the last quantifiable concentration time zero to the time of the last quantifiable concentration
Cmax | Prior to dosing（0 hour）and 0.25 hour、0.5 hour、1 hour、1.5 hours、2 hours、3 hours、4 hours、6 hours、8 hours、10 hours、12 hours、24 hours、36 hours、48 hours、72 hours、96 hours after dosing
  maximum observed plasma concentration
tmax | Prior to dosing（0 hour）and 0.25 hour、0.5 hour、1 hour、1.5 hours、2 hours、3 hours、4 hours、6 hours、8 hours、10 hours、12 hours、24 hours、36 hours、48 hours、72 hours、96 hours after dosing
  time of the maximum observed plasma concentration
t½ | Prior to dosing（0 hour）and 0.25 hour、0.5 hour、1 hour、1.5 hours、2 hours、3 hours、4 hours、6 hours、8 hours、10 hours、12 hours、24 hours、36 hours、48 hours、72 hours、96 hours after dosing
  apparent terminal elimination half-life
Vz/F | Prior to dosing（0 hour）and 0.25 hour、0.5 hour、1 hour、1.5 hours、2 hours、3 hours、4 hours、6 hours、8 hours、10 hours、12 hours、24 hours、36 hours、48 hours、72 hours、96 hours after dosing
  apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Xinghe Wang, MD, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University
Locations (1):
- Beijing shijitan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No